CLINICAL TRIAL: NCT02760043
Title: Does the Addition of Dexamethasone to a Local Infiltration Analgesia Mixture Improve Functional Outcomes Following Total Joint Arthroplasty?
Brief Title: Dexamethasone in Total Knee and Total Hip Arthroplasty
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UHN15-9898-A
Record Dates: First submitted 2016-04-14; First posted 2016-05-03 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Total Knee Arthroplasty; Total Hip Arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Dexamethasone; Calcium Dobesilate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): LIA mixture with the addition of 8mg Dexamethasone.
  Interventions: Drug: Dexamethasone; Drug: LIA Combination Mixture
- Saline (Sham Comparator): LIA mixture with the addition of 2mL of 0.9% NaCl Saline.
  Interventions: Other: 0.9% NaCl Placebo; Drug: LIA Combination Mixture

INTERVENTIONS:
Drug: Dexamethasone — 8mg (2mL) of Dexamethasone added to standard LIA mixture
  Other Names: Baycadron
  Arms: Dexamethasone
Other: 0.9% NaCl Placebo — 2mL of 0.9% NaCl placebo (saline) added to standard LIA mixture
  Other Names: Saline
  Arms: Saline
Drug: LIA Combination Mixture — 150mL 2% Ropivacaine, 30mg Ketorolac and 0.6mg of Epinephrine

SUMMARY:
This study will evaluate if the addition of dexamethasone to a local infiltration analgesia mixture will improve functional outcomes following total hip and knee arthroplasty.

DETAILED DESCRIPTION:
The addition of dexamethasone to an local infiltration analgesia (LIA) mixture for postoperative analgesia following total knee arthroplasty (TKA) has a limited evidence base. Although there is increasing support in the literature for its use in peripheral nerve blockade, there have only been a handful of studies assessing its applicability in periarticular LIA. Moreover, the evidence from peripheral nerve blocks suggests that one of the key benefits of dexamethasone is a prolongation of nerve blockade. Additionally, dexamethasone has been shown to prolong the local analgesic effect of bupivacaine microcapsules.

With respect to total hip arthroplasty (THA), there have only been two small studies that included corticosteroids in the LIA mixture; there was analgesic benefit and better early rehabilitation outcomes when compared to placebo. However, there is limited high-quality evidence for either THA or TKA demonstrating an improvement in functional outcomes when dexamethasone is used in an LIA mixture. This study will evaluate if the addition of dexamethasone to a local infiltration analgesia mixture will improve functional outcomes following total hip and knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective, primary, unilateral total hip or knee arthroplasty under spinal anesthesia
* ASA-PS I-III
* 18-85 years of age, inclusive
* 50-100 kg, inclusive
* BMI 18 - 40

Exclusion Criteria:

* Revision hip/knee arthroplasty
* Bilateral hip/knee arthroplasty
* Inability or refusal to provide informed consent
* Any contraindication to spinal anesthesia (e.g., bleeding diathesis, infection, neuropathy)
* Allergy to local anesthesia, ketorolac or dexamethasone
* Allergy to opioids
* Chronic pain state, neuropathic pain
* Opioid dependence
* Diabetic patients will NOT be excluded except those with significant peripheral neuropathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Cumulative systemic opioid consumption measured as oral morphine mg equivalents at 24 hours postoperatively | 3 days - post operative

SECONDARY OUTCOMES:
Analgesic outcomes- pain | 3 days - post operative
  Pain scores assessed with an 11 point verbal numeric rating scale (NRS) at the following time points:
  1. The post-anesthetic care unit (PACU)
  2. Postoperative day (POD) 1 at rest between 8-10 AM
  3. POD1 during physiotherapy
  4. POD 2 at rest between 8 -10 AM
  5. POD 2 during physiotherapy
  g. POD 3 during physiotherapy if still in hospital
Analgesic outcomes- opiate consumption | 3 days - post operative
  Cumulative systemic opioid consumption measured as oral morphine mg equivalents on POD 1, POD2, and, if still in hospital, POD 3, as well as the proportion of patients who required "rescue" intravenous patient controlled analgesia (IV PCA) anytime in the postoperative period
Analgesic outcomes- TUG test | 3 days - post operative
  Timed Up and Go Test (TUG) on postoperative days 2 or 3
Analgesic outcomes- Drug side-effects | 3 days - post operative
  Incidence of opioid-related side effects:
  1. Nausea and vomiting requiring treatment with anti-emetic
  2. Pruritus requiring treatment with antihistamines
  3. Sedation requiring treatment with opioid antagonist
Short-term physical and performance-based functional outcome measures- in hospital complications | 3 days post operative
  In-hospital complications- Any outcomes such as MI, surgical site infection, neurological complications, etc. that may have occurred during the hospital stay
Short-term physical and performance-based functional outcome measures- length of stay | 3 days - post operative
  Hospital length of stay- the total number of days the patient stayed in hospital to recover from elective surgery
Short-term physical and performance-based functional outcome measures- discharge | 3 days - post operatively
  Discharge destination- determination of location for which the patient was discharged; either to home or to rehabilitation centre
Medium-term self-reported functional outcome measures- WOMAC | 3 months- post operative
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measured at baseline and at 3 months post-operatively
Medium-term self-reported functional outcome measures- LFES | 3 months- post operative
  Lower extremity functional scale (LEFS) measured at baseline and at 3 months post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hopspital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this moment.

REFERENCES:
- [Derived] El-Boghdadly K, Short AJ, Gandhi R, Chan V. Addition of dexamethasone to local infiltration analgesia in elective total knee arthroplasty: double-blind, randomized control trial. Reg Anesth Pain Med. 2021 Feb;46(2):130-136. doi: 10.1136/rapm-2020-102079. Epub 2020 Nov 16. PMID 33199379
- [Derived] El-Boghdadly K, Short AJ, Gandhi R, Chan VWS. Addition of dexamethasone to local infiltration analgesia in elective total hip arthroplasty: a double-blind, randomized control trial. Reg Anesth Pain Med. 2019 Sep 27:rapm-2019-100873. doi: 10.1136/rapm-2019-100873. Online ahead of print. PMID 31563881